CLINICAL TRIAL: NCT02510248
Title: A Randomized, Double-blind, Placebo-controlled, First-in-human, 3-part Study of Orally Administered JNJ-54257099 to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Ascending Doses (Part 1) and Food-effect (Part 2) in Healthy Subjects, and Multiple Doses in Subjects With Chronic Hepatitis C Infection (Part 3)
Brief Title: First in Human Study of AL-704; Single Dose, Food Effect in Healthy Volunteers; Multiple Doses in Chronic Hepatitis C
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Alios Biopharma Inc. (Industry)
Collaborators: Janssen Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AL-704-701
Record Dates: First submitted 2015-07-02; First posted 2015-07-29 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Chronic Hepatitits C
MeSH Terms: interventions — 1-2-isopropoxy-2-oxidodihydro-4H,6H-spiro(furo(3,2-d)(1,3,2)dioxaphosphinine-7,2'-oxetan)-6-yl)pyrimidine-2,4(1H,3H)-dione

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Drug (Experimental): Study drug will be AL-704 once or twice daily for up to 7 days in dosages ranging from 100 mg to 1500 mg.
  Interventions: Drug: AL-704
- Placebo (Placebo Comparator): Placebo to match study drug dosing.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AL-704 — JNJ-54257099 (also known as ALS-022704 or AL-704) is a hepatitis C virus (HCV) nonstructural (NS)5B inhibitor, belonging to the nucleoside / nucleotide inhibitor class, and is being developed as an orally administered anti-HCV therapeutic.
  Other Names: JNJ-54257099; ALS-022704
  Arms: Study Drug
Drug: Placebo — Placebo to match AL-704
  Arms: Placebo

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, first-in-human, 3-part study in which the safety, tolerability, and pharmacokinetics of orally administered AL-704 will be assessed in healthy adult subjects and in adult subjects with CHC infection.

Part 1: Healthy adult subjects will receive one of 5 single ascending oral doses (SAD) of AL-704 ranging from 100 mg to 1,500 mg (Cohorts 1 to 5). Within each cohort subjects will be randomized to receive either AL-704 or placebo (n=8 per cohort; 6 assigned to AL-704 and 2 assigned to placebo), in a fasted state.

The planned dose-escalation scheme may be changed based on the emerging PK and safety data. Two additional cohorts (Cohorts 6 and 7) may be enrolled for evaluation of additional doses at the discretion of the Sponsor and Investigator, based on the emerging pharmacokinetic (PK) profile, and the presence of an acceptable safety profile.

Part 2: To assess the food effect on pharmacokinetics, 8 healthy subjects from one full Part 1 cohort who received a single dose of AL-704 or placebo in a fasted state, will receive the same single dose of AL-704 or placebo in a fed state in Part 2 after a washout period of 7-14 days (depending on PK results). It is expected that Cohort 3 of Part 1 (600 mg dose) will be selected, however this depends on the evaluation of available PK and safety data from Part 1 of the study.

Part 3: The following cohorts of 10 adult subjects each, with CHC infection, will be evaluated. Subjects with CHC genotype 1 infection (Cohorts 8 to 10) and subjects with CHC genotype 3 infection (Cohort 11) will be randomized to receive AL-704 or placebo for 7 consecutive days (n=10 per cohort, 8 assigned to AL-704 and 2 assigned to placebo) in a fed state. The treatment is anticipated to be administered in a once daily dose regimen or a twice daily dose regimen. The dose and dose regimen to be administered will be determined by the Sponsor depending on the PK and safety outcomes of previous cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be a man or woman 18 to 60 years of age, inclusive for healthy subjects, or 18 to 65 years of age, inclusive for subjects with CHC infection.
* Each subject must sign an ICF indicating that he or she understands the purpose of and procedures required for the study and are willing to participate in the study before starting any screening activities.
* Subject must be willing and able to adhere to the prohibitions and restrictions
* Subject included in Part 1 and 2 of the study, must be non-smokers for at least 3 months prior to screening.
* Subject included in Part 1 and 2 of the study, must be healthy on the basis of a medical evaluation that reveals the absence of any clinically relevant abnormality and includes a physical examination, medical history, vital signs, and the results of biochemistry, and hematology tests and a urinalysis performed at screening and admission. If there are abnormalities, the subject may be included only if the Investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the subject's source documents and initialed by the Investigator.
* Subject with CHC infection included in Part 3 of the study, must be otherwise healthy on the basis of a medical evaluation that reveals the absence of any clinically relevant abnormality other than those related to CHC infection, and includes a physical examination, medical history, vital signs, and the results of blood biochemistry, blood coagulation and hematology tests and a urinalysis performed at screening and admission. If there are abnormalities, the subject may be included only if the Investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the subject's source documents and initialed by the Investigator and the Sponsor.
* Subject included in Part 1 and 2 of the study, must have a body mass index (BMI) of 18.0 to 32.0 kg/m2, extremes included. Subjects with CHC infection included in Part 3 of the study must have a BMI of 18.0 to 35.0 kg/m2, extremes included, with a minimum weight of 50 kg in both populations. No more than 25% of patients in any cohort may be enrolled with a BMI ≥30 kg/m2.
* Female subject must be of non-childbearing potential.
* Female subject, except if postmenopausal, should have a negative serum pregnancy test at screening and a negative urine pregnancy test at admission.
* Subject must agree to comply with contraceptive measures .
* Subject must have a normal 12-lead ECG (based on the mean value of the triplicate parameters at admission)
* Additional inclusion criteria for CHC-infected subjects in Part 3 of the study:
* Documentation of HCV infection for longer than 6 months and determination of genotype 1 or 3 HCV infection at screening. In case of discrepancy between previously documented geno- or subtype and the geno- or subtype determined at screening, the eligibility results will be used to determine eligibility.
* HCV RNA viral load ≥105 IU/mL using a sensitive quantitative assay

Exclusion Criteria:

* Subject has a history or current clinically significant medical illness (except for
* CHC infection in subjects in Part 3 of the study) that, in the opinion of the Investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject or that could prevent, limit, or confound the protocol-specified assessments. This may include but is not limited to renal dysfunction (calculated creatinine clearance below 60 mL/min at screening), significant cardiac, vascular, pulmonary, gastrointestinal (such as significant diarrhea, gastric stasis, or constipation that in the Investigator's opinion could influence drug absorption or bioavailability), endocrine, neurologic, hematologic, rheumatologic, psychiatric, neoplastic, or metabolic disturbances.
* Subject has a positive human immunodeficiency virus type 1 or 2 (HIV-1 or HIV-2) test at screening.
* Subject has hepatitis A infection (confirmed by hepatitis A antibody immunoglobulin M [IgM]), or hepatitis B virus infection (confirmed by hepatitis B surface antigen [HBsAg]) at screening. Subject has current hepatitis C virus (HCV) infection (confirmed by HCV
* antibody) at screening, only applicable in Part 1 and 2 of the study.
* Subject has received an investigational agent (small molecule) or vaccine within 30 days, or having received a biological product within 3 months or 5 elimination half-lives (whichever is longer) prior to the planned intake of study drug.
* Subject has a past history of heart arrhythmias (extrasystole, tachycardia at rest) or of risk factors for Torsade de Pointes syndrome (eg, hypokalemia, family history of long QT Syndrome).
* Subject has donated or lost more than 1 unit of blood (500 mL) within 60 days or more than one unit of plasma within 7 days prior to the first intake of study drug.
* Subject has evidence of active infection (other than CHC infection for subjects enrolled in Part 3).
* Subject has a positive urine drug test at study screening or admission.
* Additional exclusion criteria for CHC-infected subjects in Part 3 of the study:
* Subject with HCV RNA <105 IU/mL.
* Subject has a history of clinical hepatic decompensation, eg, variceal bleeding, spontaneous bacterial peritonitis, ascites, hepatic encephalopathy or active jaundice.
* Subject has had a liver biopsy within 2 years or Fibroscan evaluation within 6 months prior to randomization that demonstrates cirrhosis (Knodell score >3, Metavir score >3, Ishak score >4). Fibroscan liver stiffness score >12.5 kPa.
* Subject has received prior treatment for CHC.
* Subject has ultrasound evidence consistent with or suspicious for hepatocellular carcinoma.
* Subject has alpha fetoprotein (AFP) >50 ng/mL, unless the absence of a hepatic mass or lesion is demonstrated by ultrasound within the screening period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-07-31 (Actual); Primary Completion 2015-11-24 (Actual); Study Completion 2015-11-24 (Actual)

PRIMARY OUTCOMES:
Safety Data assessed by Number and frequency of treatment emergent adverse events, physical examination findings | From screening to last visit (up to 21 days)
  abnormal vital signs, 12 lead ECG and abnormal clinical laboratory results examination findings, vital signs, ECG and clinical lab results

SECONDARY OUTCOMES:
Single dose PK Profile from Cmax, tmax, t1/2, CL/F and Vz/F, AUC0-inf or AUClast | From dosing to Day 8 visit for each SAD/FE cohort
Multiple dose PK: profile from Cmax, tmax, t1/2, AUClast and AUC0 tau | From dosing to final study visit (21 days) for each cohort
Hepatitis C virus levels | From screening to final study visit (21 days) for each cohort
  HCV RNA viral load change from baseline to final study visit in subjects with Chronic hepatitis C infection

CONTACTS AND LOCATIONS:
Locations (3):
- Biotrial, Rennes, Brittany Region, France
- Arensia, Tbilisi, Georgia
- Arensia, Chisinau, Moldova